CLINICAL TRIAL: NCT00750867
Title: Treatment of Multiple System Atrophy Using Intravenous Immunoglobulins
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Peter Novak, Study Principle Investigator, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-12784
Record Dates: First submitted 2008-09-09; First posted 2008-09-11 (Estimated); Results first posted 2015-10-26 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2015-09

CONDITIONS: Multiple System Atrophy
Keywords: multiple system atrophy, MSA,; intravenous immunoglobulin, IVIg
MeSH Terms: conditions — Multiple System Atrophy; Thyroid Dyshormonogenesis 2A | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Interventions included monthly infusions of intravenous immunoglobulin.
  Interventions: Drug: intravenous immunoglobulin (IVIg)

INTERVENTIONS:
Drug: intravenous immunoglobulin (IVIg) — The intravenous immunoglobulin (brand Privigen) will be infused intravenously, monthly, 6 times, for 6 months the dose will be 0.4 gram/kg for each infusion.
  Other Names: Privigen

SUMMARY:
Multiple System Atrophy (MSA) is a progressive sporadic neurodegenerative disorder leading to widespread loss of brain cells that results in parkinsonian, cerebellar and autonomic dysfunction. The cause of the MSA remains unclear. Available treatment is symptomatic only and does not alter the course of disease.

Although the cause of MSA remains unclear, there is evidence of presence of common neuroinflammatory mechanisms in the MSA brains including activation of microglia and production of toxic cytokines. This research protocol is based on hypothesis that the MSA progression can be altered by blocking the neuroinflammatory activity.

This protocol includes administration of intravenous immunoglobulin (IVIg). IVIg contains antibodies derived from human plasma which can block the inflammatory responses in the brain that can lead to loss of brain cells.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female older than 17 years.
2. Clinical diagnosis of probable multiple system atrophy
3. Provide written informed consent to participate in the study
4. Understand that they may withdraw their consent at any time

Exclusion Criteria:

1. Women who are pregnant or lactating
2. In the investigator's opinion, have any other significant systemic, hepatic, cardiac or renal illness.
3. In the investigator's opinion, the subjects are significantly dehydrated, as determined by clinical evaluation including measurement of skin turgor, blood urea nitrogen and creatinine values.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Novak, MD, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Result] Novak P, Williams A, Ravin P, Zurkiya O, Abduljalil A, Novak V. Treatment of multiple system atrophy using intravenous immunoglobulin. BMC Neurol. 2012 Nov 1;12:131. doi: 10.1186/1471-2377-12-131. PMID 23116538

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Interventional Arm: intravenous immunoglobulin (IVIg): The IVIg will be infused intravenously, monthly, 6 times, the dose will be 0.4 gram/kg for each infusion.
Period: Overall Study
Arm/Group | Open Label Interventional Arm
Started | 9
Completed | 7
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Interventional Arm
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 59 [55 to 64]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events up to Six Months Post-treatment
Description: The primary outcome measure was to evaluate the safety and tolerability of the IVIG infusions in patients with multiple system atrophy. The primary endpoint was defined as the frequency of adverse events (AE). AEs including their severity and relationship to the IVIG were assessed throughout the study and at least 60 days after the last infusion. The AEs were considered to be related to the IVIG infusion (infusional AE) if they occurred during an infusion or within 72 hours afterwards. Non-infusional AEs were further classified as possible related to IVIG or likely not related to IVIG. Serious AEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization. Any AE was defined as occurrence of any symptom regardless of intensity grade.
Time Frame: Monthly, up to 8 months (including the screening visit and the final visit)
Population: Two participants dropped out from the study.
Measure: Number; unit: Adverse events
Arm/Group | Open Label Interventional Arm
Number analyzed (Participants) | 7
Adverse events
  All Adverse Events | 43
  Serious Adverse Events | 0

2. Secondary Outcome: Preliminary Efficacy of IVIg for Treatment of MSA.
Description: The secondary outcome measure was to evaluate the preliminary efficacy of IVIG for the treatment of MSA. The primary efficacy endpoint was change of the Unified MSA Rating Scale (UMSARS-I and UMSAR-II) compared to baseline. UMSARS-I and UMSARS-II are validated semiquantitative rating scales for evaluation of severity of MSA. UMSARS-I comprises a historical review of disease-related impairments and UMSARS-II comprises motor examination. UMSARS-I has 12 questions, each with assigned score 0-4, where 0 is normal and > are abnormal responses. Total range of UMSARS-I is 0 to 48. UMSARS-II has 12 items rated by an examiner, each with assigned score 0-4, where 0 is normal and > are abnormal responses. Total range of UMSARS-II is 0 to 56. The scores of UMSARS-I and UMSARS-II at baseline (month 1) was compared with the scores obtained at the final visit (month 8) which was 8 months apart. The interventions occured at months 2-7, total six times.
Time Frame: Monthly, up to 8 months (including the screening visit and the final visit)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label Interventional Arm
Number analyzed (Participants) | 7
units on a scale
  UMSARS-I, baseline | 23.8 (6)
  UMSARS-II,baseline | 26.1 (7.4)
  UMSARS-I, final visit | 19 (5.9)
  UMSARS-II, final visit | 23.3 (7.2)
Statistical Analysis 1: Comparison: Open Label Interventional Arm; Test type: Superiority or Other; p = 0.0128, ANOVA — The P-Value was obtained by comparing the UMSARS-I scores at final visit and at baseline
Statistical Analysis 2: Comparison: Open Label Interventional Arm; Test type: Superiority or Other; p = 0.025, ANOVA — The P-Value was obtained by comparing the UMSARS-II scores at final visit and at baseline

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Open Label Interventional Arm
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Interventional Arm (N=9)
elevated blood pressure (Vascular disorders) | 9 (32) — transient, responding to adjusting the infusion rate
urinary tract infection (Infections and infestations) | 1 (1) — treated with antibiotics
Accidental injury (Respiratory, thoracic and mediastinal disorders) | 1 (1) — nose fracture
pruritic skin rash (Skin and subcutaneous tissue disorders) | 3 (4) — 2 subjects withdrew from the study.
increased temperature or skin flushing (Skin and subcutaneous tissue disorders) | 1 (5) — treated with Diphenhydramine, Acetaminophen, and slowing the infusion rate
restless leg syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) — treated with iron supplements
decreased GFR (Renal and urinary disorders) | 2 (2) — resolved
ankle edema (Vascular disorders) | 1 (1) — treated with diuretics
elevated BUN (Renal and urinary disorders) | 1 (1) — resolved
worsening of allergies (Skin and subcutaneous tissue disorders) | 2 (2)
nodular lung abnormality (Respiratory, thoracic and mediastinal disorders) | 1 (1) — later determined to be a tangle of vein most likely inborn
low potassium (Endocrine disorders) | 1 (1) — treated with potassium supplements
viral infection of gastrointenstinal tract (Gastrointestinal disorders) | 1 (1) — resolved
elevated PSA (Reproductive system and breast disorders) | 1 (1) — resolved
wrist strain (Musculoskeletal and connective tissue disorders) | 1 (1) — resolved
worsening of sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — treated with continuous positive airway pressure (CPAP)

LIMITATIONS AND CAVEATS:
The main study limitation is its small size and open label character.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No